CLINICAL TRIAL: NCT03321877
Title: Down-titration of Steroids in Patients With Difficult Asthma With no Bronchial Hyperreactivity: Severe Asthma or Simply Over-treatment?
Brief Title: Down-titration of Steroids in Patients With Difficult Asthma With no Bronchial Hyperreactivity
Acronym: DOSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Eileen Wedge, Research doctor, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 55855
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All included patients underwent dose reduction.
  Interventions: Drug: Change to dose of patient's regular medication

INTERVENTIONS:
Drug: Change to dose of patient's regular medication — Dose reduction of the drug each patient was already taking

SUMMARY:
An 8 week 'real-life' inhaled corticosteroid (ICS) dose reduction study in patients with severe asthma without evidence of bronchial hyperactivity.

DETAILED DESCRIPTION:
We aim to describe the proportion of patients with severe asthma, but without objective evidence of active disease, who can successfully be reduced in ICS dose for a period of 8 weeks. This is also intended as an exploration of the methodology and feasibility of step-down studies with this patient group, to act as a pilot for future projects.

This study enrolled patients from the SATS severe asthma study, in which they had undergone systematic investigation for comorbidities, triggers and barriers to good asthma control.

After baseline investigations, the patient's ICS dose is halved (or as close as possible to, but not below, 50%). Patients continued on the same inhaled steroid drug and device. Patients taking a combined ICS/LABA inhaler halve the dose of this, as per usual clinical practice. Other asthma medicaitons are continued unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma for at least 6 months
* Fulfill ERS/ATS giudelines for severe asthma
* Stable dose of ICS for at least 4 weeks
* Able to carry out study procedures
* Negative metacholine provocation test at screening
* Negative reversibility to beta agonist at screening
* FeNO under 50 ppb

Exclusion Criteria:

* Treatment with prednisolone, methotrexate, ciclosporin, omalizumab or nucala in the last 6 months
* FEV1 under 70% of predicted
* Acute upper or lower airway infection requiring antibiotics in the last 4 weeks
* Exacerbation of asthma requiring prednisolone in the last 6 months
* Current smoking
* Pregnancy or breastfeeding
* Other clinically significant lung disease
* Current participation in another interventional study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Responsiveness to metacholine bronchial challenge | 8 weeks
  PD(20) if positive test

SECONDARY OUTCOMES:
ACQ score | 8 weeks
  asthma control questionnaire
miniAQLQ score | 8 weeks
  asthma quality of life score
Pulmonary function tests | 8 weeks
  FEV1, FVC, reversibility to beta agonist
FeNO | 8 weeks
  fraction of exhaled nitric oxide
Sputum cell differentials | 8 weeks
  sputum neutrophil and eosinophil counts

CONTACTS AND LOCATIONS:
Locations (1):
- Lungemedicinsk Forskningsenhed, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No